CLINICAL TRIAL: NCT02299193
Title: Online CBT-I for High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Faye Routledge, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00073066
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Hypertension; Prehypertension; Insomnia
Keywords: cognitive behavioral therapy for insomnia; sleep hygiene
MeSH Terms: conditions — Hypertension; Prehypertension; Sleep Initiation and Maintenance Disorders; Sleep Hygiene | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): online sessions on how behaviors and thoughts that can affect sleep.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Healthy Sleep Habits (Sham Comparator): online sessions about healthy sleep practices
  Interventions: Behavioral: Healthy Sleep Habits

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 6 weekly, 20 minute online sessions about how thoughts and behaviors can affect sleep
  Other Names: CBT-I
  Arms: Cognitive Behavioral Therapy
Behavioral: Healthy Sleep Habits — 6 weekly, 20 minute online sessions about healthy sleep practices
  Arms: Healthy Sleep Habits

SUMMARY:
The purpose of this study is to compare the effect of 6-weekly, 20 minute sessions of 2 online behavioral sleep interventions (cognitive behavioral therapy or healthy sleep habits) on blood pressure, sleep, depressive symptoms and anxiety in people with insomnia and prehypertension or hypertension.

DETAILED DESCRIPTION:
Approximately 30% of US adults have prehypertension (untreated blood pressure ≥120-139/80-89 mmHg) and 29% have hypertension (blood pressure ≥ 140/90 mmHg or antihypertensive medication use). Numerous factors contribute to the development of prehypertension and hypertension including age, genetics, obesity, and behavioral factors such as exercise and diet.However, the sleep disorder insomnia is another behavioral factor increasingly implicated with risk of hypertension. Insomnia, the most frequent sleep complaint in adults, is characterized by difficulty falling asleep, trouble maintaining sleep or non-restorative sleep coupled with significant daytime distress or functional impairment. Insomnia is a pervasive sleep disorder associated with decreased quality of life, reduced work productivity, and increased health care costs; it is increasingly identified as a cardiovascular disease risk factor. Lifestyle modifications recommended for pre-hypertension and hypertension do not address sleep. This pilot randomized clinical trial will test the preliminary efficacy of an online cognitive behavioral therapy intervention (N=40) versus an online healthy sleep habits intervention (N=20), to reduce blood pressure in a sample of untreated individuals with insomnia and prehypertension or hypertension. Participants will be followed for 12-weeks post-intervention. Primary outcome measures are systolic blood pressure. Secondary measures include sleep efficiency, insomnia severity, physical and mental function.

ELIGIBILITY:
Inclusion Criteria:

* prehypertension or hypertension, insomnia (difficulty getting to sleep, staying asleep and/or early morning awakenings), internet access, current email use, willingness to be randomized to either intervention group, ability to read/write in English.

Exclusion Criteria:

* medication known to alter sleep, sleep disorder (other than insomnia), frequent travel over 2-3 time zones, currently receiving behavioral treatment for insomnia, major depression, anxiety disorders, PTSD or bipolar disorder, >14 alcoholic drinks/week, recreational drug use, prior diagnosis of: epilepsy, dementia/Alzheimer's disease, renal failure requiring dialysis, stroke, secondary hypertension, angina, peripheral artery disease, heart failure, myocardial infarction or cardiac surgery within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | 8 and 20 weeks
  Systolic blood pressure will be measured at baseline, 8 and 20 weeks

SECONDARY OUTCOMES:
Change in Insomnia Severity Index | 8 and 20 weeks
  Insomnia Severity Index (ISI) questionnaire will be measured at baseline, 8 and 20 weeks
Changes in Sleep Efficiency | 8 and 20 weeks
  Actigraphy based sleep efficiency will be measured at baseline, 8 and 20 weeks
Change in Depressive Symptoms | 8 and 20 weeks
  Depressive symptoms measured at baseline, 8 and 20 weeks
Change in mental functioning | 8 and 20 weeks
  Mental function measured at baseline, 8 and 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States